CLINICAL TRIAL: NCT00613782
Title: Testosterone Replacement Therapy in Men With Type 2 Diabetes Mellitus and Low Testosterone Levels
Brief Title: Reandron in Diabetic Men Witn Low Testosterone Level
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Austin Health (Other Government)
Responsible Party: Principal Investigator, Mathis Grossmann, AProf, Austin Health
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Reandron 1000 (ZK 5488) 321399
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2012-06

CONDITIONS: Type 2 Diabetes; Hypogonadism
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypogonadism | interventions — testosterone undecanoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Reandron 100 treatment
  Interventions: Drug: Reandron 1000
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Reandron 1000 — 1000mg at 0,6,18,30 weeks
  Other Names: testosterone undecanoate
  Arms: 1
Drug: placebo — placebo injection 0,6.18.30 weeks
  Arms: 2

SUMMARY:
In men with type 2 diabetes, low testosterone levels have been associated with insulin resistance, truncal obesity and symptoms such as fatigue and erectile dysfunction. Low testosterone may impair cardiac function and increase cardiovascular risk and cause osteoporosis. The goal of this project is to assess prospectively whether, in men with type 2 diabetes mellitus and low testosterone levels, testosterone replacement improves insulin resistance, body composition, bone density, cardiac function symptoms associated with low testosterone level.

The investigators will recruit 140 ambulatory men with type 2 diabetes and a low serum testosterone level (<10 nmol/L) from Austin Health Endocrine clinics, General Practise surgeries, and from the general public by direct consumer advertising via newspaper and other local media. Men will be randomised to either intramuscular testosterone undecanoate (Reandron 1000, Bayer Schering Pharma) or placebo. Men with contraindications to testosterone replacement or to intramuscular injections will be excluded from the study. All men will receive intramuscular testosterone or placebo injections at 0, 6, 18 and 30 weeks (a total of four injections).

All 140 study subjects will have a clinical and laboratory assessment at baseline, 18 weeks and at study end (40 weeks). All 140 subjects will also have imaging studies at baseline and at study end (40 weeks). The study protocol is outlined in more detail below:

Clinical and laboratory assessment (Baseline and repeated 18 weeks, 40 weeks) A full medical history and physical examination will be performed. Symptoms will be assessed by the following standardised questionnaires: 1) Androgen Deficiency in the Aging Male (ADAM); 2) Aging Male Symptom scale (AMS); 3) International Index of Erectile Dysfunction (IIED); 4) International Prostate Symptom Score (IPSS); 5) SF-36 (all five questionnaires are attached to Module 1).

Laboratory studies will consist of blood tests to measure total testosterone, fasting glucose, C-peptide, HBA1c and other routine parameters.

Imaging studies (Baseline and repeated at 40 weeks)

1. Body composition and bone mineral density by DEXA
2. Body composition by magnetic resonance imaging
3. Bony micro-architecture by high resolution quantitative computed tomography [HR-pQCT]),
4. Cardiac dimensions and function by transthoracic doppler echocardiography

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Testosterone less than 10 nmol/L

Exclusion Criteria:

* Contraindication to
* Testosterone or
* IM injection

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2009-01; Primary Completion 2014-01 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Insulin Resistance | 40 weeks

SECONDARY OUTCOMES:
Bone microarchitecture | 40 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mathis Grossmann, Principal Investigator — Austin Health
Locations (1):
- Austin Health, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Gianatti EJ, Dupuis P, Hoermann R, Zajac JD, Grossmann M. Effect of testosterone treatment on constitutional and sexual symptoms in men with type 2 diabetes in a randomized, placebo-controlled clinical trial. J Clin Endocrinol Metab. 2014 Oct;99(10):3821-8. doi: 10.1210/jc.2014-1872. Epub 2014 Jun 30. PMID 24978674